CLINICAL TRIAL: NCT04502459
Title: A Prospective Randomized Trial on the Use of Tourniquet in Primary Total Knee Arthroplasty
Brief Title: A Study on the Use of Tourniquet Use In Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yan Chun-Hoi, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW 15-129
Record Dates: First submitted 2020-07-14; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Osteo Arthritis Knee; Rheumatoid Arthritis of Knee
Keywords: Tourniquet; Total Knee Arthroplasty
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: A randomization list was generated prior to recruitment using a computer software (Random Allocation Software Version 1.0.0, Isfahan, Iran). The participants were randomly allocated to either of the 3 groups with different tourniquet strategies: Group 1) tourniquet inflation from skin to cement hardening (skin to cement); Group 2) tourniquet inflation only from cementation (cement only); Group 3) tourniquet inflation from skin incision to skin closure (skin to skin). The surgeon opened a sealed envelope containing the allocation right before the operation in the theatre. The evaluators who examined and collected the data were blinded to the patients' allocation to the study groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cement only (Active Comparator): The tourniquet was inﬂated just before cement application and deﬂated after its hardening
  Interventions: Procedure: Tourniquet
- Skin to Cement (Active Comparator): Inﬂation of tourniquet before skin incision and its deﬂation after hardening of cement
  Interventions: Procedure: Tourniquet
- Skin to Skin (Active Comparator): Inflate of tourniquet before incision and deflate following completion of skin closure
  Interventions: Procedure: Tourniquet

INTERVENTIONS:
Procedure: Tourniquet — A tourniquet is often used in total knee arthroplasty to achieve better visualization, reduce intra-operative bleeding and facilitate cement interdigitation

SUMMARY:
A tourniquet is often used in total knee arthroplasty (TKA) to achieve better visualization, reduce intra-operative bleeding and facilitate cement interdigitation. On the other hand, the associated risks include skin burns, soft tissue and muscle damage, injury of calcified vessels, increased swelling and stiffness of the joints, nerve injury, paralysis, and thromboembolic events. The automatic lower limb pneumatic tourniquet system (Zimmer) was applied to reduce blood loss during surgery. A prospective randomized controlled trial (RCT) was performed to investigate the best tourniquet strategy in TKA. The participants were randomly allocated to groups with different tourniquet strategies: Group 1) tourniquet inflation from skin to cement hardening (skin to cement); Group 2) tourniquet inflation only from cementation (cement only) and Group 3) tourniquet inflation from skin incision to skin closure (skin to skin). In addition to the blood loss and early postoperative outcomes, pain, soft tissue injury, and rehabilitation were also strictly monitored with a longer follow-up duration up to 6 months.

DETAILED DESCRIPTION:
A tourniquet is often used in total knee arthroplasty (TKA) to achieve better visualization, reduce intra-operative bleeding and facilitate cement interdigitation. On the other hand, the associated risks include skin burns, soft tissue and muscle damage, injury of calcified vessels, increased swelling and stiffness of the joints, nerve injury, paralysis, and thromboembolic events.

The automatic lower limb pneumatic tourniquet system (Zimmer) was applied to reduce blood loss during surgery. The skin under the tourniquet was covered by cast padding. The operated leg was elevated and exsanguinated before inﬂating the automatic pneumatic tourniquet. There are three main strategies for the use of a tourniquet in TKR: A) inflate before incision and deflate following cement hardening ('skin to cement'); B) inflate prior to cement application and deflated following hardening ('cement only'); C) inflate before incision and deflate following completion of skin closure ('skin to skin'). The optimal timing of tourniquet application during primary TKA is still a matter of debate. Most previous reports have failed to show signiﬁcant differences among different tourniquet strategies.

Kvederas et al. compared these three strategies in a randomized double-blind clinical trial, and demonstrated that the estimated blood loss was highest when the tourniquet was inﬂated just before cement application and deﬂated after its hardening ('cement only'), while inﬂation of tourniquet before skin incision and its deﬂation after hardening of cement ('skin to cement') tends to give better early postoperative mobilization. However, this was an interim report with limited number of patients, and only limited outcome parameters were reported, which were insufﬁcient to draw ﬁrm conclusions regarding the differences in outcome.

Therefore we performed this prospective randomized controlled trial (RCT) with a decent sample size to investigate the best tourniquet strategy in TKA. In addition to the blood loss and early postoperative outcomes, we also strictly monitored pain, soft tissue injury, and rehabilitation with a longer follow-up duration up to 6 months.

All of the operations were performed through the medial parapatellar approach by the same experienced joint replacement surgeon. All patients underwent primary TKA with minimally invasive techniques and cemented prostheses (EvolutionTM medial pivot, MicroPort, USA). An intramedullary guide was used for both tibial and femoral cuts.

The automatic lower limb pneumatic tourniquet system was applied to reduce blood loss during surgery. The skin under the tourniquet was covered by cast padding. The operated leg was elevated and exsanguinated before inﬂating the automatic pneumatic tourniquet. One of the three tourniquet treatment strategies was used, as determined by the group allocation of the patient. In all the three groups, the tourniquet was inﬂated to a pressure of 280 mm Hg. The wound was closed after wound irrigation and hemostasis and then was wrapped with elastic bandages. One drainage was applied postoperatively in all patients and was kept until 24h to monitor blood loss.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffer from primary osteoarthritis indicated for total knee arthroplasty
2. Subject is physically and mentally willing and able to comply with the postoperative scheduled clinical and radiographic evaluations
3. Subject must have signed an informed consent document specific to the study, and approved by the Ethics Committee, indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

1. Subject requires a revision knee arthroplasty surgery
2. Subject is currently on anti-coagulant therapy or has coagulopathy
3. Subject has peripheral vascular disease of the lower limb evidenced by the presence of blood vessel calcification on the radiographs or the absence of dorsalis pedis/popliteal pulses
4. Subject suffers from conditions other than primary knee osteoarthritis, e.g. inflammatory arthritis
5. Subject having associated medical diseases affecting rehabilitation
6. Subject has active systemic infection or infection near the knee joint
7. Subject having current medical condition that render them unfit for surgery
8. Any criterion which in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Blood Loss | 4 days after surgery
  We calculated the intraoperative blood loss by measuring the suction volume and weighing the sponges. Hemoglobin (Hb) and hematocrit (Hct) levels were examined preoperatively, and on Day 1 to Day 4 after surgery. Change of Hb and Hct was calculated as the value of postoperative D1 to D4 minus preoperative value. The number of patients undergoing blood transfusion were recorded. The criterion for a blood transfusion was set as a Hb level of <8 g/dL with symptomatic anemia. The calculated blood loss, which reﬂects actual blood loss, was determined with use of a previously described method. Briefly, the patients blood volume (PBV) is calculated using a formula, and multiplying the PBV by the change of haematocrit (preoperative value minus value on postoperative Day 2) will give the estimated total blood loss (ETBL).

SECONDARY OUTCOMES:
Soft-tissue damage | 4 days after surgery
  We assessed soft-tissue damage by examining serum C-reactive protein (CRP), creatine kinase (CK), lactate dehydrogenase (LDH), and interleukin-6 (IL-6) levels preoperatively and on postoperative days 1, 2, 3 and 4
Thigh circumference | 4 days after surgery
  Thigh circumference was measured 10 cm proximal to the patella and leg circumference was measured 15 cm distal to the patella, to determine the degree of swelling, and was measured on postoperative days 1, 2, 3 and 4. X-rays were taken after surgery to measure the lower limb alignment, and tibial and femoral components position.
Postoperative Visual Analog Scale | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  Postoperative visual analog scale (VAS) scores were obtained for both knee and thigh pain preoperatively and on postoperative.
Peak Quadriceps Strength | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  The strength of each leg was evaluated by using an isokinetic dynamometer. Peak torque measured in both the concentric and eccentric modes.
Time-up-and-go (TUG) Test | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  he TUG test was used to evaluate the preoperative degree of mobility. This test involves measuring the time a patient needs to get up from a chair, walk three meters, turn, walk back to the chair and then sit down again.
6-minute Walking Test | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  A test that evaluates the functional capacity of the patient while walking on a flat, hard surface in the 6-minute window. It assess all the systems that are involved in the 6-minute window.
Berg Balance Scale | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  The BBS test is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Knee Society Knee Score | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  A knee score that rates only the knee joint itself, there are three main parameters which are pain, stability and the range of motion. Whereas flexion contracture, extension lag and misalignment would be different ways for point deductions. 100 points would refer to a patient with no knee pain, 125 degree range of motion and negligible anteroposterior and mediolateral instability.
Knee Society Function Score | Day 1, Day 2, Day 3, Day 4, Day 7, Week 6, Month 3, and Month 6
  A functional score that rates the patient's ability to walk and climb stairs, points would be deducted if the patient uses any walking aids for the two. 100 points would refer to a patient that can walk for an unlimited distance and go up and down the stairs without any trouble.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tai TW, Chang CW, Lai KA, Lin CJ, Yang CY. Effects of tourniquet use on blood loss and soft-tissue damage in total knee arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2012 Dec 19;94(24):2209-15. doi: 10.2106/JBJS.K.00813. PMID 23318610
- [Background] Tarwala R, Dorr LD, Gilbert PK, Wan Z, Long WT. Tourniquet use during cementation only during total knee arthroplasty: a randomized trial. Clin Orthop Relat Res. 2014 Jan;472(1):169-74. doi: 10.1007/s11999-013-3124-2. PMID 23836239